CLINICAL TRIAL: NCT05060965
Title: Smoking Cessation Pilot Program on 9 South
Brief Title: Inpatient Smoking Cessation Pilot Program
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No Enrollees
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00208192
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cessation intervention (Experimental): All participants will receive nicotine replacement therapy and a referral to both Maryland Quitline and Johns Hopkins Tobacco Treatment Clinic for continued cessation care.
  Nicotine replacement therapy: Nicoderm patches, gum, lozenges
  * Low nicotine dependence: Lozenge (2 mg) or Gum (2 mg) or Patch (7 mg)
  * Moderate nicotine dependence: Patch (14 mg) and Lozenge (2 mg) or Gum (2 mg)
  * High nicotine dependence: Patch (21 mg) and Lozenge (4 mg) or Gum (4 mg)
  Regardless of the level of nicotine addiction and subsequent dose of nicotine replacement therapy (NRT), participants of this trials are described as "recipients of NRT products".
  Interventions: Drug: Nicotine lozenge; Drug: Nicotine gum; Drug: Nicotine patch; Other: Maryland Quitline; Other: John Hopkins Tobacco Treatment Clinic

INTERVENTIONS:
Drug: Nicotine lozenge — Nicotine replacement therapy
Drug: Nicotine gum — Nicotine replacement therapy
Drug: Nicotine patch — Nicotine replacement therapy
Other: Maryland Quitline — Telephone-based tobacco cessation service
Other: John Hopkins Tobacco Treatment Clinic — Clinic-based tobacco cessation service

SUMMARY:
The investigators are implementing a stepwise approach to cessation with a public health focus to improve health outcomes for the investigators' pediatric patients. The investigators are focusing on addressing caregiver smoking as a modifiable risk factor during time of child's hospitalization as a window of opportunity to provide counseling and education to families on secondhand and third hand smoke exposure as well as information on NRT products to heighten caregiver contemplation for quitting. One of the central goals of the investigators' project is to increase immediate access to Nicotine Replacement Therapy (NRT) resources for families during hospitalization which pediatric providers could potentially dose and prescribe to caregivers who are screened positive for smoking. Long-term cessation care is provided by referrals to both the MD Quitline and the John Hopkins Tobacco Treatment Clinic. Both are provided to allow participants options that the participants would find preferable from an insurance and provider perspective.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients on an inpatient unit at Johns Hopkins Children's Center who self-identify as tobacco users and wish to initiate tobacco cessation

Exclusion Criteria:

* Pregnant or breast feeding maternal caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Self-reported attempts to quit smoking | Baseline, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months
  Change in caregiver self-reported tobacco cessation attempt in the past 14-days.

SECONDARY OUTCOMES:
Change in Frequency of usage of outpatient tobacco cessation services | Baseline, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months
  Change in frequency of caregiver self-reported usage of outpatient tobacco cessation services (Maryland Quitline or Johns Hopkins Tobacco Treatment Clinic).
Change in Usage of nicotine replacement therapy products | Baseline, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months
  Change in caregiver self-reported usage of nicotine replacement therapy in the past 14-days.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep S. Jassal, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data will be shared with researchers or sponsor upon review of a written request. The request will require a detailed description of the usage of the data and will require approval by the principal investigator. A data use agreement will be set-up and a plan for data removal (including timeline) will be established.